CLINICAL TRIAL: NCT00600821
Title: Randomized Phase 2 Trial Of AG013736 Or Bevacizumab In Combination With Paclitaxel And Carboplatin As First Line Treatment For Patients With Advanced Non Small Cell Lung Cancer
Brief Title: A Study Of AG-013736 (Axitinib) Or Bevacizumab (Avastin) In Combination With Paclitaxel And Carboplatin In Patients With Advanced Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4061030
Record Dates: First submitted 2008-01-03; First posted 2008-01-25 (Estimated); Results first posted 2012-05-22 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Non-Small-Cell Lung Carcinoma; Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma | interventions — Bevacizumab; Carboplatin; Paclitaxel; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator): Bevacizumab will be administered in combination with carboplatin and paclitaxel.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel
- A (Experimental): AG-013736 will be administered in combination with carboplatin and paclitaxel.
  Interventions: Drug: AG-013736 (axitinib); Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is available as 100 and 400 mg preservative-free, single use vials- The starting dose is 15 mg/kg, iv infusion, every 3 weeks.
  Other Names: Avastin
  Arms: B
Drug: Carboplatin — Carboplatin is available as pre-mixed 10mg /ml aqueous solution- The starting dose is AUC 6 mg*min/ml, iv infusion, every 3 weeks.
  Arms: B
Drug: Paclitaxel — Paclitaxel is available in multidose vials (30 mg/5ml;100mg/16.7 ml;300 mg/50ml)- The starting dose is 200 mg/m2, every 3 weeks
  Arms: B
Drug: AG-013736 (axitinib) — AG-013736 (axitinib) is available as 1mg, and 5 mg film-coated tablets for oral administration- The starting dose is 5 mg BID-
  Other Names: axitinib Taxol
  Arms: A
Drug: Carboplatin — Carboplatin is available as pre-mixed 10mg /ml aqueous solution- The starting dose is AUC 6 mg*min/ml, iv infusion, every 3 weeks.
  Arms: A
Drug: Paclitaxel — Paclitaxel is available in multidose vials (30 mg/5ml;100mg/16.7 ml;300 mg/50ml)- The starting dose is 200 mg/m2, every 3 weeks
  Arms: A

SUMMARY:
To determine if the addition of AG-013736 to chemotherapy is beneficial in patients with advanced lung cancer who have not been previously treated.

ELIGIBILITY:
Inclusion Criteria:

* Advanced non squamous cell, lung cancer
* No prior treatment for lung cancer except prior adjuvant therapy if last dose was >12 months prior to enrollment

Exclusion Criteria:

* Prior therapy for advanced lung cancer
* The need for blood-thinners
* Coughing up blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (17):
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Columbus, Mississippi
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, New Albany, Mississippi
  - Pfizer Investigational Site, Oxford, Mississippi
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Bartlett, Tennessee
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Lubbock, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Wenatchee, Washington
- Czechia (3):
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Tábor
  - Pfizer Investigational Site, Ústí nad Labem
- France (3):
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pierre-Bénite
- Poland (5):
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Gdynia
  - Pfizer Investigational Site, Torun
  - Pfizer Investigational Site, Warsaw
- Spain (4):
  - Pfizer Investigational Site, Alicante, Alicante
  - Pfizer Investigational Site, Mataró, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Valencia, Valencia
- United Kingdom (6):
  - Pfizer Investigational Site, Southampton, Hampshire
  - Pfizer Investigational Site, Dundee, Scotland
  - Pfizer Investigational Site, Leeds, Yorkshire
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Surrey

REFERENCES:
- [Derived] Twelves C, Chmielowska E, Havel L, Popat S, Swieboda-Sadlej A, Sawrycki P, Bycott P, Ingrosso A, Kim S, Williams JA, Chen C, Olszanski AJ, de Besi P, Schiller JH. Randomised phase II study of axitinib or bevacizumab combined with paclitaxel/carboplatin as first-line therapy for patients with advanced non-small-cell lung cancer. Ann Oncol. 2014 Jan;25(1):132-8. doi: 10.1093/annonc/mdt489. PMID 24356624
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061030&StudyName=A%20Study%20Of%20AG-013736%20%28Axitinib%29%20Or%20Bevacizumab%20%28Avastin%29%20In%20Combination%20With%20Paclitaxel%20And%20Carboplatin%20In%20Patients%20With%20Advanced%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib + Paclitaxel + Carboplatin: Axitinib (AG-013736) 5 milligram (mg) tablet administered orally twice daily (BID) along with infusion of paclitaxel 200 mg per square meter (mg/m^2) over 3 hours and carboplatin area under the concentration-time curve (AUC) of 6 mg*minute/milliliter (mg*min/mL) infusion over 30 minutes in cycles of 3 weeks. After completion or discontinuation of treatment for reasons other than disease progression, participants continued to receive axitinib (AG-013736) BID maintenance therapy.
- Bevacizumab + Paclitaxel + Carboplatin: Bevacizumab 15 mg/kilogram (mg/kg) infusion over 90 minutes every 3 weeks along with infusion of paclitaxel 200 mg/m^2 over 3 hours and carboplatin AUC of 6 mg*min/mL infusion over 30 minutes in cycles of 3 weeks. After completion or discontinuation of treatment for reasons other than disease progression, participants continued to receive bevacizumab maintenance therapy every 3 weeks.
Period: Overall Study
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Started | 58 | 60
Treated | 58 | 59
Completed | 0 | 0
Not Completed | 58 | 60
Not completed — Death | 45 | 46
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Terminated by sponsor | 8 | 6
Not completed — Objective progression or relapse | 0 | 1
Not completed — Randomized but not treated | 0 | 1
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug, or received a different drug from that to which they were randomized.
Groups:
- Axitinib + Paclitaxel + Carboplatin: Axitinib (AG-013736) 5 mg tablet administered orally BID along with IV infusion of paclitaxel 200 mg per square meter (mg/m^2) over 3 hours and carboplatin AUC of 6 mg*min/mL infusion over 30 minutes in cycles of 3 weeks. After completion or discontinuation of treatment for reasons other than disease progression, participants continued to receive axitinib (AG-013736) BID maintenance therapy.
- Bevacizumab + Paclitaxel + Carboplatin: Bevacizumab 15 mg/kg infusion over 90 minutes every 3 weeks along with infusion of paclitaxel 200 mg/m^2 over 3 hours and carboplatin AUC of 6 mg*min/mL infusion over 30 minutes in cycles of 3 weeks. After completion or discontinuation of treatment for reasons other than disease progression, participants continued to receive bevacizumab maintenance therapy every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Customized [Number; unit: Participants]
  Less than 18 years | 0 | 0 | 0
  18 to 44 years | 1 | 2 | 3
  45 to 64 years | 33 | 44 | 77
  Greater than or equal to 65 years | 24 | 14 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time in months from start of study treatment to first randomization date of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the first randomization date plus 1) divided by 30.4. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline, every 6 weeks until disease progression or initiation of subsequent anticancer therapy up to 2.75 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 58 | 60
Months | 5.7 [4.1 to 7.5] | 6.1 [4.2 to 8.7]
Statistical Analysis 1: Comparison: Axitinib + Paclitaxel + Carboplatin vs Bevacizumab + Paclitaxel + Carboplatin; Differences in PFS between treatment arms was analyzed by 1-sided log rank test, stratified by gender and prior adjuvant therapy; Test type: Superiority or Other; p = 0.639, Log Rank — One-sided log-rank test at alpha = 0.20 significance level was used; Hazard Ratio (HR) = 1.093, 95% CI 2-sided [0.679 to 1.761]

2. Secondary Outcome: Overall Survival (OS)
Description: Time in months from date of randomization to date of death due to any cause. OS was calculated as (the death date minus the first randomization date plus 1) divided by 30.4. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline, every 6 weeks until death or bimonthly after final study visit (up to 2.75 years)
Population: ITT population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug, or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 58 | 60
Months | 10.6 [7.5 to 16.4] | 13.3 [10.4 to 17.6]
Statistical Analysis 1: Comparison: Axitinib + Paclitaxel + Carboplatin vs Bevacizumab + Paclitaxel + Carboplatin; Differences in OS between treatment arms was analyzed by 1-sided log rank test, stratified by gender and prior adjuvant therapy; Test type: Superiority or Other; p = 0.699, Log Rank — One-sided log-rank test at alpha = 0.20 significance level was used; Hazard Ratio (HR) = 1.117, 95% CI 2-sided [0.739 to 1.689]

3. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed response were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. CR: disappearance of all lesions (target and/or non target) and no appearance of new lesions. PR: at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, without progression of non target lesions and no appearance of new lesions.
Time Frame: Baseline, every 6 weeks until disease progression or initiation of subsequent anticancer therapy up to 2.75 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 58 | 60
Percentage of participants | 29.3 [18.1 to 42.7] | 43.3 [30.6 to 56.8]
Statistical Analysis 1: Comparison: Axitinib + Paclitaxel + Carboplatin vs Bevacizumab + Paclitaxel + Carboplatin; P-value was calculated using 1-sided Cochran-Mantel-Haenszel test stratified by gender and prior adjuvant therapy. Risk ratio in comparison to the Bevacizumab group was calculated assuming all other factors as constant; Test type: Superiority or Other; p = 0.9422, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.676, 95% CI 2-sided [0.412 to 1.107]

4. Secondary Outcome: Duration of Response (DR)
Description: Time in months from the first documentation of objective tumor response that is subsequently confirmed to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to any cause minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.4. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Baseline, every 6 weeks until disease progression or initiation of subsequent anticancer therapy up to 2.75 years
Population: DR was calculated for the subgroup of participants from the ITT population, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 17 | 26
Months | 4.4 [4.2 to 6.7] | 7.0 [4.8 to 8.3]

5. Secondary Outcome: Population Pharmacokinetic (PK) Analysis for Axitinib (AG-013736)
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Pre-dose, 1 to 2 hours post-dose on Cycle 2 of Day 1 and Cycle 3 of Day 1
Reporting Status: Not Posted

6. Secondary Outcome: European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhoea, and financial difficulties). Most questions used 4- point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Time Frame: Day (D) 1 of every cycle (C) then every 3 weeks until final study visit (up to 2.75 years)
Population: ITT population included participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or different drug from which they were randomized. 'n' signifies those participants evaluated for this measure at specific time point for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 58 | 60
Units on a scale
  Physical functioning (PF): Baseline (n=58, 59) | 66.29 (22.04) | 75.00 (22.21)
  PF: C2 D1 (n=51, 53) | 67.45 (23.48) | 75.47 (20.24)
  PF: C3 D1 (n=45, 47) | 65.78 (24.40) | 78.16 (18.43)
  PF: C4 D1 (n=37, 48) | 67.88 (20.01) | 73.78 (19.14)
  PF: C5 D1 (n=34, 38) | 61.18 (24.09) | 75.09 (16.38)
  PF: C6 D1 (n=31, 33) | 65.86 (19.17) | 73.94 (18.66)
  PF: C7 D1 (n=27, 30) | 66.42 (22.15) | 74.89 (18.67)
  PF: C8 D1 (n=22, 28) | 67.27 (22.44) | 77.14 (18.98)
  PF: C9 D1 (n=18, 23) | 66.30 (27.77) | 74.57 (19.02)
  PF: C10 D1 (n=17, 20) | 68.63 (25.36) | 81.33 (14.92)
  PF: C11 D1 (n=15, 19) | 60.67 (23.58) | 78.25 (16.00)
  PF: C12 D1 (n=10, 17) | 71.33 (20.86) | 78.43 (19.65)
  PF: C13 D1 (n=8, 14) | 66.67 (25.94) | 79.05 (21.22)
  PF: End of treatment (EOT) (n=27, 38) | 62.96 (21.11) | 64.91 (24.83)
  Role functioning: Baseline (n=58, 58) | 60.92 (31.15) | 60.63 (31.79)
  Role functioning: C2 D1 (n=51, 53) | 64.38 (31.98) | 65.41 (29.02)
  Role functioning: C3 D1 (n=45, 47) | 58.15 (34.01) | 70.92 (28.55)
  Role functioning: C4 D1 (n=37, 48) | 67.12 (26.49) | 67.36 (25.02)
  Role functioning: C5 D1 (n=34, 38) | 57.35 (29.64) | 66.23 (29.12)
  Role functioning: C6 D1 (n=31, 33) | 62.90 (30.34) | 67.68 (29.15)
  Role functioning: C7 D1 (n=28, 30) | 55.36 (32.41) | 63.89 (27.01)
  Role functioning: C8 D1 (n=22, 28) | 65.15 (29.05) | 71.43 (19.70)
  Role functioning: C9 D1 (n=18, 23) | 63.89 (37.60) | 70.29 (18.77)
  Role functioning: C10 D1 (n=17, 20) | 66.67 (28.87) | 70.83 (20.14)
  Role functioning: C11 D1 (n=15, 19) | 60.00 (29.41) | 71.93 (21.55)
  Role functioning: C12 D1 (n=10, 17) | 75.00 (21.15) | 70.59 (21.67)
  Role functioning: C13 D1 (n=8, 14) | 62.50 (33.04) | 80.95 (20.52)
  Role functioning: EOT (n=27, 38) | 57.41 (32.47) | 57.90 (31.18)
  Emotional functioning: Baseline (n=57, 57) | 69.74 (23.45) | 63.74 (27.44)
  Emotional functioning: C2 D1 (n=50, 53) | 78.33 (21.76) | 73.64 (22.81)
  Emotional functioning: C3 D1 (n=45, 48) | 75.19 (21.36) | 78.76 (20.69)
  Emotional functioning: C4 D1 (n=37, 48) | 75.75 (20.17) | 76.04 (23.23)
  Emotional functioning: C5 D1 (n=32, 38) | 77.60 (18.38) | 78.51 (21.37)
  Emotional functioning: C6 D1 (n=29, 32) | 78.74 (18.97) | 77.35 (23.40)
  Emotional functioning: C7 D1 (n=28, 30) | 78.57 (22.62) | 79.45 (20.50)
  Emotional functioning: C8 D1 (n=22, 28) | 77.65 (19.14) | 81.25 (18.09)
  Emotional functioning: C9 D1 (n=18, 23) | 74.07 (19.78) | 78.50 (23.39)
  Emotional functioning: C10 D1 (n=17, 20) | 77.94 (18.85) | 78.33 (13.36)
  Emotional functioning: C11 D1 (n=15, 19) | 70.00 (21.32) | 82.46 (18.61)
  Emotional functioning: C12 D1 (n=10, 17) | 74.17 (27.90) | 77.45 (20.57)
  Emotional functioning: C13 D1 (n=8, 14) | 77.08 (22.60) | 83.93 (14.79)
  Emotional functioning: EOT (n=27, 38) | 68.52 (26.39) | 70.18 (25.60)
  Cognitive Functioning: Baseline (n=57, 57) | 80.12 (24.28) | 83.33 (19.16)
  Cognitive Functioning: C2 D1 (n=50, 53) | 84.00 (20.47) | 84.28 (21.29)
  Cognitive Functioning: C3 D1 (n=45, 48) | 85.19 (22.81) | 85.42 (20.81)
  Cognitive Functioning: C4 D1 (n=37, 48) | 84.68 (18.99) | 82.64 (20.03)
  Cognitive Functioning: C5 D1 (n=32, 38) | 84.37 (19.83) | 83.33 (24.51)
  Cognitive Functioning: C6 D1 (n=29, 32) | 86.78 (18.03) | 81.25 (21.06)
  Cognitive Functioning: C7 D1 (n=28, 30) | 79.76 (19.43) | 85.56 (18.94)
  Cognitive Functioning: C8 D1 (n=22, 28) | 89.39 (17.48) | 88.69 (17.00)
  Cognitive Functioning: C9 D1 (n=18, 23) | 84.26 (15.63) | 86.23 (20.51)
  Cognitive Functioning: C10 D1 (n=17, 20) | 88.23 (12.86) | 90.00 (13.68)
  Cognitive Functioning: C11 D1 (n=15, 19) | 82.22 (18.33) | 85.96 (18.64)
  Cognitive Functioning: C12 D1 (n=10, 17) | 90.00 (14.05) | 87.25 (20.01)
  Cognitive Functioning: C13 D1 (n=8, 14) | 85.42 (13.91) | 95.24 (12.10)
  Cognitive Functioning: EOT (n=27, 38) | 77.78 (23.57) | 78.95 (22.82)
  Social functioning: Baseline (n=57, 57) | 71.35 (27.59) | 65.50 (32.25)
  Social functioning: C2 D1 (n=50, 52) | 69.67 (30.06) | 75.32 (25.24)
  Social functioning: C3 D1 (n=45, 48) | 71.11 (27.62) | 74.65 (24.79)
  Social functioning: C4 D1 (n=37, 48) | 73.42 (24.99) | 71.53 (29.77)
  Social functioning: C5 D1 (n=32, 38) | 65.10 (26.22) | 75.88 (27.04)
  Social functioning: C6 D1 (n=29, 32) | 70.11 (26.49) | 71.88 (26.92)
  Social functioning: C7 D1 (n=28, 30) | 64.88 (32.50) | 72.22 (23.71)
  Social functioning: C8 D1 (n=22, 28) | 71.97 (24.87) | 72.02 (24.45)
  Social functioning: C9 D1 (n=18, 23) | 74.07 (29.83) | 81.16 (16.13)
  Social functioning: C10 D1 (n=17, 20) | 72.55 (32.24) | 79.17 (20.14)
  Social functioning: C11 D1 (n=15, 19) | 66.67 (28.17) | 78.95 (16.52)
  Social functioning: C12 D1 (n=10, 17) | 71.67 (20.86) | 80.39 (20.61)
  Social functioning: C13 D1 (n=8, 14) | 56.25 (28.08) | 80.95 (18.32)
  Social functioning: EOT (n=27, 38) | 69.14 (26.03) | 65.79 (26.83)
  Fatigue: Baseline (n=57, 58) | 40.45 (23.94) | 38.89 (28.02)
  Fatigue: C2 D1 (n=51, 53) | 43.57 (21.98) | 36.48 (25.26)
  Fatigue: C3 D1 (n=45, 47) | 47.41 (22.77) | 33.80 (19.38)
  Fatigue: C4 D1 (n=37, 48) | 42.34 (19.22) | 37.85 (19.40)
  Fatigue: C5 D1 (n=34, 38) | 44.61 (21.73) | 36.84 (22.83)
  Fatigue: C6 D1 (n=31, 33) | 45.16 (23.65) | 33.50 (21.45)
  Fatigue: C7 D1 (n=28, 30) | 47.82 (27.27) | 40.74 (21.11)
  Fatigue: C8 D1 (n=22, 28) | 44.95 (24.84) | 32.14 (20.14)
  Fatigue: C9 D1 (n=18, 23) | 40.12 (29.80) | 28.98 (20.03)
  Fatigue: C10 D1 (n=17, 20) | 41.83 (25.62) | 30.00 (19.78)
  Fatigue: C11 D1 (n=15, 19) | 47.78 (32.52) | 28.07 (14.52)
  Fatigue: C12 D1 (n=10, 17) | 37.78 (19.74) | 29.41 (18.82)
  Fatigue: C13 D1 (n=8, 14) | 50.00 (24.49) | 26.19 (22.05)
  Fatigue: EOT (n=27, 38) | 51.03 (24.51) | 43.13 (27.57)
  Nausea and vomiting: Baseline (n=57, 59) | 8.77 (17.85) | 9.89 (21.91)
  Nausea and vomiting: C2 D1 (n=51, 53) | 7.19 (13.02) | 5.35 (12.56)
  Nausea and vomiting: C3 D1 (n=45, 47) | 11.11 (17.77) | 5.67 (11.67)
  Nausea and vomiting: C4 D1 (n=37, 48) | 10.81 (16.77) | 7.29 (11.86)
  Nausea and vomiting: C5 D1 (n=34, 38) | 13.24 (21.63) | 7.46 (14.34)
  Nausea and vomiting: C6 D1 (n=31, 33) | 13.44 (21.26) | 10.61 (17.59)
  Nausea and vomiting: C7 D1 (n=28, 30) | 15.48 (22.65) | 9.44 (14.31)
  Nausea and vomiting: C8 D1 (n=22, 28) | 14.40 (22.00) | 5.95 (12.18)
  Nausea and vomiting: C9 D1 (n=18, 23) | 9.26 (13.06) | 5.07 (20.98)
  Nausea and vomiting: C10 D1 (n=17, 20) | 11.77 (15.33) | 8.33 (16.67)
  Nausea and vomiting: C11 D1 (n=15, 19) | 14.45 (17.67) | 5.26 (9.71)
  Nausea and vomiting: C12 D1 (n=10, 17) | 15.00 (16.57) | 6.68 (14.50)
  Nausea and vomiting: C13 D1 (n=8, 14) | 12.50 (17.25) | 5.95 (14.03)
  Nausea and vomiting: EOT (n=27, 38) | 16.05 (22.40) | 7.90 (14.36)
  Pain: Baseline (n=57, 59) | 31.29 (31.82) | 35.31 (30.02)
  Pain: C2 D1 (n=51, 53) | 29.74 (29.87) | 28.30 (29.16)
  Pain: C3 D1 (n=45, 48) | 30.00 (27.43) | 18.75 (18.07)
  Pain: C4 D1 (n=37, 48) | 26.58 (18.62) | 25.35 (27.29)
  Pain: C5 D1 (n=34, 38) | 25.00 (18.91) | 24.12 (24.72)
  Pain: C6 D1 (n=31, 33) | 31.18 (18.63) | 25.25 (28.90)
  Pain: C7 D1 (n=28, 30) | 28.57 (28.99) | 27.22 (26.07)
  Pain: C8 D1 (n=22, 28) | 28.03 (25.91) | 22.62 (23.66)
  Pain: C9 D1 (n=18, 23) | 33.33 (22.14) | 27.54 (31.22)
  Pain: C10 D1 (n=17, 20) | 30.39 (26.51) | 24.17 (24.47)
  Pain: C11 D1 (n=15, 19) | 43.33 (28.03) | 18.42 (21.44)
  Pain: C12 D1 (n=10, 17) | 35.00 (21.45) | 23.53 (29.50)
  Pain: C13 D1 (n=8, 14) | 35.42 (24.30) | 16.67 (21.68)
  Pain: EOT (n=27, 38) | 38.27 (33.27) | 34.65 (30.36)
  Dyspnoea: Baseline (n=56, 58) | 32.74 (30.15) | 36.21 (33.21)
  Dyspnoea: C2 D1 (n=51, 52) | 32.03 (28.25) | 24.36 (31.04)
  Dyspnoea: C3 D1 (n=45, 47) | 38.52 (28.39) | 19.15 (23.82)
  Dyspnoea: C4 D1 (n=37, 48) | 33.33 (30.43) | 21.53 (25.25)
  Dyspnoea: C5 D1 (n=34, 38) | 36.27 (33.20) | 23.68 (27.84)
  Dyspnoea: C6 D1 (n=31, 33) | 36.56 (31.45) | 20.20 (23.48)
  Dyspnoea: C7 D1 (n=28, 30) | 38.09 (31.05) | 21.11 (20.50)
  Dyspnoea: C8 D1 (n=22, 28) | 27.27 (28.43) | 16.67 (19.24)
  Dyspnoea: C9 D1 (n=18, 23) | 25.93 (33.44) | 21.74 (21.58)
  Dyspnoea: C10 D1 (n=17, 20) | 27.45 (31.70) | 18.33 (17.01)
  Dyspnoea: C11 D1 (n=15, 19) | 37.78 (33.01) | 17.54 (23.22)
  Dyspnoea: C12 D1 (n=10, 17) | 23.33 (27.44) | 21.57 (23.40)
  Dyspnoea: C13 D1 (n=8, 14) | 37.50 (37.53) | 19.05 (17.12)
  Dyspnoea: EOT (n=27, 38) | 35.80 (27.62) | 33.33 (33.78)
  Insomnia: Baseline (n=57, 58) | 46.20 (33.19) | 37.93 (31.50)
  Insomnia: C2 D1 (n=51, 53) | 36.60 (36.06) | 28.30 (33.59)
  Insomnia: C3 D1 (n=45, 47) | 30.37 (33.20) | 29.08 (33.06)
  Insomnia: C4 D1 (n=37, 48) | 24.32 (26.81) | 27.08 (28.89)
  Insomnia: C5 D1 (n=34, 38) | 28.43 (24.80) | 23.68 (31.87)
  Insomnia: C6 D1 (n=31, 33) | 24.73 (25.77) | 24.24 (29.19)
  Insomnia: C7 D1 (n=28, 30) | 23.81 (28.48) | 25.55 (24.26)
  Insomnia: C8 D1 (n=22, 28) | 21.21 (26.32) | 19.05 (23.00)
  Insomnia: C9 D1 (n=18, 23) | 25.93 (31.43) | 23.19 (27.40)
  Insomnia: C10 D1 (n=17, 20) | 27.45 (26.97) | 20.00 (25.13)
  Insomnia: C11 D1 (n=15, 19) | 33.33 (28.17) | 22.81 (24.97)
  Insomnia: C12 D1 (n=10, 17) | 26.67 (21.08) | 23.53 (28.30)
  Insomnia: C13 D1 (n=8, 14) | 12.50 (17.25) | 16.67 (17.29)
  Insomnia: EOT (n=27, 37) | 28.39 (27.28) | 36.94 (30.21)
  Loss of appetite: Baseline (n=57, 59) | 29.82 (28.65) | 31.64 (34.14)
  Loss of appetite: C2 D1 (n=51, 53) | 23.53 (26.91) | 20.75 (29.40)
  Loss of appetite: C3 D1 (n=44, 47) | 33.33 (32.94) | 17.02 (25.89)
  Loss of appetite: C4 D1 (n=37, 48) | 26.13 (26.22) | 23.61 (27.47)
  Loss of appetite: C5 D1 (n=34, 38) | 30.39 (33.20) | 21.05 (29.43)
  Loss of appetite: C6 D1 (n=31, 33) | 27.96 (31.15) | 23.23 (26.98)
  Loss of appetite: C7 D1 (n=28, 30) | 39.29 (34.01) | 24.44 (23.05)
  Loss of appetite: C8 D1 (n=22, 28) | 36.36 (28.93) | 19.05 (21.14)
  Loss of appetite: C9 D1 (n=18, 23) | 31.48 (26.75) | 13.04 (24.08)
  Loss of appetite: C10 D1 (n=17, 20) | 39.22 (31.70) | 20.00 (25.13)
  Loss of appetite: C11 D1 (n=15, 19) | 33.33 (35.64) | 15.79 (17.10)
  Loss of appetite: C12 D1 (n=10, 17) | 16.67 (23.57) | 23.53 (30.65)
  Loss of appetite: C13 D1 (n=8, 14) | 29.17 (21.36) | 16.67 (28.49)
  Loss of appetite: EOT (n=27, 38) | 39.51 (34.64) | 37.72 (33.93)
  Constipation: Baseline (n=56, 57) | 15.48 (23.75) | 21.05 (31.89)
  Constipation: C2 D1 (n=50, 53) | 21.33 (28.38) | 20.13 (26.43)
  Constipation: C3 D1 (n=45, 47) | 18.52 (24.16) | 14.89 (23.88)
  Constipation: C4 D1 (n=36, 48) | 18.52 (26.96) | 13.19 (21.46)
  Constipation: C5 D1 (n=32, 38) | 18.75 (22.30) | 21.05 (27.31)
  Constipation: C6 D1 (n=28, 33) | 22.62 (25.75) | 19.19 (28.90)
  Constipation: C7 D1 (n=28, 30) | 25.00 (26.64) | 7.78 (14.34)
  Constipation: C8 D1 (n=22, 28) | 19.70 (19.68) | 2.38 (8.74)
  Constipation: C9 D1 (n=18, 23) | 9.26 (19.15) | 5.80 (12.92)
  Constipation: C10 D1 (n=17, 20) | 17.65 (20.81) | 5.00 (12.21)
  Constipation: C11 D1 (n=15, 19) | 22.22 (20.57) | 8.77 (18.73)
  Constipation: C12 D1 (n=10, 17) | 20.00 (23.31) | 5.88 (17.62)
  Constipation: C13 D1 (n=8, 14) | 16.67 (25.20) | 4.76 (12.10)
  Constipation: EOT (n=27, 38) | 20.99 (29.45) | 14.03 (24.05)
  Diarrhoea: Baseline (n=55, 57) | 6.67 (17.45) | 5.85 (14.26)
  Diarrhoea: C2 D1 (n=50, 53) | 11.33 (17.31) | 10.06 (21.27)
  Diarrhoea: C3 D1 (n=45, 48) | 15.55 (18.26) | 9.72 (21.70)
  Diarrhoea: C4 D1 (n=37, 47) | 13.51 (19.97) | 5.67 (12.66)
  Diarrhoea: C5 D1 (n=32, 38) | 22.92 (32.17) | 7.89 (18.07)
  Diarrhoea: C6 D1 (n=29, 32) | 21.84 (28.56) | 10.42 (19.74)
  Diarrhoea: C7 D1 (n=28, 30) | 16.67 (26.45) | 11.11 (15.98)
  Diarrhoea: C8 D1 (n=22, 28) | 24.24 (31.17) | 4.76 (11.88)
  Diarrhoea: C9 D1 (n=18, 23) | 27.78 (28.58) | 5.80 (12.92)
  Diarrhoea: C10 D1 (n=17, 20) | 23.53 (30.65) | 10.00 (19.04)
  Diarrhoea: C11 D1 (n=15, 19) | 31.11 (34.43) | 0.00 (0.00)
  Diarrhoea: C12 D1 (n=10, 17) | 43.33 (16.10) | 0.00 (0.00)
  Diarrhoea: C13 D1 (n=8, 14) | 33.33 (25.20) | 7.14 (14.19)
  Diarrhoea: EOT (n=27, 38) | 23.46 (28.96) | 3.51 (12.94)
  Financial difficulties: Baseline (n=56, 57) | 22.62 (31.85) | 21.64 (27.09)
  Financial difficulties: C2 D1 (n=49, 53) | 21.77 (31.59) | 20.12 (27.22)
  Financial difficulties: C3 D1 (n=45, 48) | 25.93 (30.89) | 18.05 (23.78)
  Financial difficulties: C4 D1 (n=37, 48) | 21.62 (27.46) | 20.83 (30.46)
  Financial difficulties: C5 D1 (n=32, 38) | 26.04 (30.21) | 21.05 (28.39)
  Financial difficulties: C6 D1 (n=29, 32) | 26.44 (28.70) | 20.83 (29.02)
  Financial difficulties: C7 D1 (n=28, 30) | 26.19 (31.89) | 26.67 (30.83)
  Financial difficulties: C8 D1 (n=21, 28) | 28.57 (35.41) | 21.43 (32.98)
  Financial difficulties: C9 D1 (n=18, 23) | 27.78 (36.60) | 17.39 (29.93)
  Financial difficulties: C10 D1 (n=17, 19) | 27.45 (33.82) | 24.56 (33.04)
  Financial difficulties: C11 D1 (n=15, 19) | 20.00 (30.34) | 19.30 (27.92)
  Financial difficulties: C12 D1 (n=10, 17) | 13.33 (23.31) | 17.65 (26.66)
  Financial difficulties: C13 D1 (n=8, 14) | 20.83 (35.36) | 16.67 (28.49)
  Financial difficulties: EOT (n=27, 37) | 23.46 (27.45) | 28.83 (32.55)
  Global health status/QoL: Baseline (n=57, 57) | 53.22 (22.03) | 54.97 (21.06)
  Global health status/QoL: C2 D1 (n=49, 53) | 58.16 (20.38) | 59.59 (17.78)
  Global health status/QoL: C3 D1 (n=45, 48) | 56.67 (20.07) | 59.72 (16.34)
  Global health status/QoL: C4 D1 (n=37, 47) | 57.21 (18.02) | 57.80 (18.17)
  Global health status/QoL: C5 D1 (n=32, 38) | 58.07 (21.94) | 61.84 (17.61)
  Global health status/QoL: C6 D1 (n=29, 32) | 53.45 (17.75) | 60.94 (17.51)
  Global health status/QoL: C7 D1 (n=28, 30) | 55.65 (20.17) | 58.61 (15.39)
  Global health status/QoL: C8 D1 (n=22, 28) | 56.82 (17.18) | 60.71 (15.36)
  Global health status/QoL: C9 D1 (n=18, 22) | 56.48 (23.14) | 64.40 (15.89)
  Global health status/QoL: C10 D1 (n=17, 20) | 55.39 (17.91) | 62.50 (14.93)
  Global health status/QoL: C11 D1 (n=15, 19) | 47.78 (19.02) | 63.60 (15.52)
  Global health status/QoL: C12 D1 (n=10, 17) | 54.17 (19.35) | 63.73 (12.48)
  Global health status/QoL: C13 D1 (n=8, 14) | 53.13 (19.89) | 58.33 (15.68)
  Global health status/QoL: EOT (n=27, 38) | 49.38 (20.92) | 50.22 (21.62)

7. Secondary Outcome: European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire Lung Cancer-13 (QLQ- LC13) Score
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The 13 questions comprised 1 multi-item scale for dyspnoea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, other pain, and medicine for pain). Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: Day 1 of every cycle then every 3 weeks until final study visit (up to 2.75 years)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 58 | 60
Units on a scale
  Cough: Baseline (n=56, 59) | 37.50 (31.18) | 38.42 (24.62)
  Cough: C2 D1 (n=50, 53) | 30.67 (24.13) | 30.19 (20.94)
  Cough: C3 D1 (n=46, 47) | 28.98 (25.92) | 28.37 (23.03)
  Cough: C4 D1 (n=37, 48) | 29.73 (25.80) | 27.08 (20.23)
  Cough: C5 D1 (n=33, 38) | 22.22 (18.00) | 28.07 (23.92)
  Cough: C6 D1 (n=29, 33) | 26.44 (24.20) | 26.26 (23.21)
  Cough: C7 D1 (n=28, 29) | 25.00 (21.52) | 25.29 (24.65)
  Cough: C8 D1 (n=22, 27) | 21.21 (19.37) | 19.75 (21.20)
  Cough: C9 D1 (n=18, 23) | 20.37 (20.26) | 24.64 (25.06)
  Cough: C10 D1 (n=17, 20) | 23.53 (25.73) | 21.67 (22.36)
  Cough: C11 D1 (n=15, 19) | 24.44 (23.46) | 26.31 (23.78)
  Cough: C12 D1 (n=10, 17) | 26.66 (14.05) | 29.41 (30.92)
  Cough: C13 D1 (n=8, 14) | 33.33 (25.20) | 21.43 (21.11)
  Cough: End of treatment (EOT) (n=26, 38) | 33.33 (21.08) | 33.33 (29.00)
  Haemoptysis: Baseline (n=56, 59) | 2.98 (11.51) | 3.39 (10.16)
  Haemoptysis: C2 D1 (n=50, 53) | 2.67 (9.13) | 1.89 (7.78)
  Haemoptysis: C3 D1 (n=44, 47) | 0.76 (5.02) | 5.67 (14.44)
  Haemoptysis: C4 D1 (n=36, 48) | 0.93 (5.56) | 3.47 (10.29)
  Haemoptysis: C5 D1 (n=33, 38) | 1.01 (5.80) | 3.51 (12.94)
  Haemoptysis: C6 D1 (n=29, 33) | 3.45 (13.64) | 3.03 (12.81)
  Haemoptysis: C7 D1 (n=27, 29) | 0.00 (0.00) | 3.45 (10.33)
  Haemoptysis: C8 D1 (n=22, 27) | 0.00 (0.00) | 1.23 (6.41)
  Haemoptysis: C9 D1 (n=18, 23) | 0.00 (0.00) | 0.00 (0.00)
  Haemoptysis: C10 D1 (n=17, 20) | 0.00 (0.00) | 0.00 (0.00)
  Haemoptysis: C11 D1 (n=15, 19) | 0.00 (0.00) | 0.00 (0.00)
  Haemoptysis: C12 D1 (n=10, 17) | 0.00 (0.00) | 0.00 (0.00)
  Haemoptysis: C13 D1 (n=8, 14) | 4.17 (11.78) | 0.00 (0.00)
  Haemoptysis: EOT (n=26, 38) | 0.00 (0.00) | 5.26 (16.49)
  Dyspnoea: Baseline (n=56, 58) | 29.17 (20.60) | 31.42 (28.85)
  Dyspnoea: C2 D1 (n=48, 53) | 29.86 (25.23) | 23.90 (21.51)
  Dyspnoea: C3 D1 (n=45, 43) | 33.83 (22.09) | 20.41 (18.61)
  Dyspnoea: C4 D1 (n=36, 45) | 32.10 (20.01) | 24.69 (21.57)
  Dyspnoea: C5 D1 (n=33, 37) | 30.30 (21.21) | 23.12 (19.84)
  Dyspnoea: C6 D1 (n=28, 31) | 35.32 (24.76) | 21.86 (18.70)
  Dyspnoea: C7 D1 (n=27, 27) | 30.45 (25.52) | 20.16 (16.02)
  Dyspnoea: C8 D1 (n=22, 26) | 24.75 (21.94) | 21.37 (16.61)
  Dyspnoea: C9 D1 (n=18, 22) | 27.78 (29.83) | 18.69 (14.70)
  Dyspnoea: C10 D1 (n=17, 19) | 28.76 (27.80) | 19.88 (15.08)
  Dyspnoea: C11 D1 (n=15, 18) | 27.41 (24.80) | 19.75 (15.51)
  Dyspnoea: C12 D1 (n=10, 17) | 23.33 (22.50) | 22.22 (19.25)
  Dyspnoea: C13 D1 (n=8, 14) | 37.50 (31.95) | 16.67 (16.16)
  Dyspnoea: EOT (n=25, 37) | 34.22 (23.33) | 33.63 (28.39)
  Sore Mouth: Baseline (n=56, 58) | 3.57 (12.19) | 1.15 (6.13)
  Sore Mouth: C2 D1 (n=51, 53) | 18.95 (26.88) | 9.43 (23.00)
  Sore Mouth: C3 D1 (n=45, 47) | 18.52 (28.03) | 9.22 (21.65)
  Sore Mouth: C4 D1 (n=37, 48) | 21.62 (31.64) | 8.33 (21.19)
  Sore Mouth: C5 D1 (n=33, 38) | 23.23 (36.79) | 11.40 (23.60)
  Sore Mouth: C6 D1 (n=28, 33) | 16.67 (30.77) | 6.06 (19.46)
  Sore Mouth: C7 D1 (n=28, 29) | 17.86 (27.94) | 6.90 (16.38)
  Sore Mouth: C8 D1 (n=22, 27) | 16.67 (30.43) | 3.70 (10.67)
  Sore Mouth: C9 D1 (n=18, 23) | 9.26 (15.36) | 5.80 (16.37)
  Sore Mouth: C10 D1 (n=17, 20) | 19.61 (33.46) | 10.00 (26.71)
  Sore Mouth: C11 D1 (n=15, 19) | 22.22 (37.09) | 8.77 (24.45)
  Sore Mouth: C12 D1 (n=10, 17) | 16.67 (23.57) | 7.84 (18.74)
  Sore Mouth: C13 D1 (n=8, 14) | 25.00 (38.83) | 4.76 (12.10)
  Sore Mouth: EOT (n=26, 38) | 8.97 (24.14) | 4.39 (13.80)
  Dysphagia: Baseline (n=56, 59) | 6.55 (17.31) | 6.78 (14.88)
  Dysphagia: C2 D1 (n=51, 53) | 11.76 (22.92) | 6.92 (17.73)
  Dysphagia: C3 D1 (n=46, 47) | 13.77 (20.58) | 4.96 (11.99)
  Dysphagia: C4 D1 (n=37, 48) | 9.91 (20.59) | 2.78 (9.31)
  Dysphagia: C5 D1 (n=32, 38) | 12.50 (26.44) | 4.39 (11.42)
  Dysphagia: C6 D1 (n=28, 33) | 13.10 (27.73) | 7.07 (16.15)
  Dysphagia: C7 D1 (n=28, 28) | 11.90 (26.00) | 5.95 (15.85)
  Dysphagia: C8 D1 (n=22, 27) | 16.67 (26.73) | 1.23 (6.41)
  Dysphagia: C9 D1 (n=18, 23) | 9.26 (15.36) | 1.45 (6.95)
  Dysphagia: C10 D1 (n=17, 20) | 21.57 (26.20) | 6.67 (17.44)
  Dysphagia: C11 D1 (n=15, 19) | 24.44 (29.46) | 1.75 (7.65)
  Dysphagia: C12 D1 (n=10, 17) | 6.67 (14.05) | 3.92 (16.17)
  Dysphagia: C13 D1 (n=8, 14) | 20.83 (24.80) | 4.76 (17.82)
  Dysphagia: EOT (n=26, 38) | 7.69 (21.72) | 7.89 (19.66)
  Peripheral neuropathy: Baseline (n=56, 59) | 9.52 (19.81) | 15.25 (26.50)
  Peripheral neuropathy: C2 D1 (n=51, 53) | 24.84 (30.44) | 33.96 (33.01)
  Peripheral neuropathy: C3 D1 (n=46, 47) | 37.68 (34.15) | 34.75 (36.09)
  Peripheral neuropathy: C4 D1 (n=37, 48) | 45.05 (37.86) | 38.19 (32.97)
  Peripheral neuropathy: C5 D1 (n=33, 38) | 50.51 (39.19) | 42.11 (33.50)
  Peripheral neuropathy: C6 D1 (n=29, 33) | 55.17 (39.11) | 52.53 (33.37)
  Peripheral neuropathy: C7 D1 (n=28, 29) | 48.81 (37.93) | 54.02 (33.82)
  Peripheral neuropathy: C8 D1 (n=22, 27) | 57.58 (40.08) | 50.62 (36.25)
  Peripheral neuropathy: C9 D1 (n=17, 23) | 45.10 (40.73) | 56.52 (36.84)
  Peripheral neuropathy: C10 D1 (n=17, 20) | 45.10 (42.40) | 48.33 (38.20)
  Peripheral neuropathy: C11 D1 (n=14, 19) | 50.00 (42.87) | 49.12 (35.78)
  Peripheral neuropathy: C12 D1 (n=9, 17) | 55.56 (40.83) | 54.90 (38.98)
  Peripheral neuropathy: C13 D1 (n=8, 14) | 58.33 (42.73) | 47.62 (38.60)
  Peripheral neuropathy: EOT (n=25, 38) | 37.33 (35.12) | 40.35 (38.87)
  Alopecia: Baseline (n=56, 59) | 2.98 (11.51) | 2.26 (10.48)
  Alopecia: C2 D1 (n=50, 53) | 69.33 (33.56) | 71.70 (32.29)
  Alopecia: C3 D1 (n=46, 45) | 73.91 (37.13) | 68.89 (38.53)
  Alopecia: C4 D1 (n=37, 45) | 65.77 (40.43) | 60.00 (42.40)
  Alopecia: C5 D1 (n=33, 35) | 61.62 (44.19) | 64.76 (44.24)
  Alopecia: C6 D1 (n=28, 32) | 69.05 (42.48) | 61.46 (45.68)
  Alopecia: C7 D1 (n=28, 28) | 39.29 (46.31) | 40.48 (45.68)
  Alopecia: C8 D1 (n=21, 27) | 42.86 (44.90) | 44.44 (48.92)
  Alopecia: C9 D1 (n=18, 23) | 27.78 (43.16) | 31.88 (44.36)
  Alopecia: C10 D1 (n=17, 20) | 31.37 (43.25) | 11.67 (29.17)
  Alopecia: C11 D1 (n=14, 18) | 16.67 (36.40) | 16.67 (34.77)
  Alopecia: C12 D1 (n=10, 17) | 13.33 (28.11) | 9.80 (28.30)
  Alopecia: C13 D1 (n=8, 14) | 8.33 (23.57) | 7.14 (26.73)
  Alopecia: EOT (n=26, 37) | 33.33 (42.16) | 27.03 (39.94)
  Chest pain: Baseline (n=56, 59) | 23.81 (28.93) | 20.90 (25.45)
  Chest pain: C2 D1 (n=51, 53) | 18.95 (27.69) | 10.06 (18.00)
  Chest pain: C3 D1 (n=45, 47) | 14.81 (25.18) | 5.67 (12.66)
  Chest pain: C4 D1 (n=36, 48) | 14.81 (24.49) | 9.03 (19.13)
  Chest pain: C5 D1 (n=33, 38) | 11.11 (19.84) | 3.51 (10.37)
  Chest pain: C6 D1 (n=28, 33) | 15.48 (21.24) | 1.01 (5.80)
  Chest pain: C7 D1 (n=28, 28) | 11.90 (18.62) | 3.57 (10.50)
  Chest pain: C8 D1 (n=22, 27) | 13.64 (16.77) | 3.70 (10.67)
  Chest pain: C9 D1 (n=18, 23) | 12.96 (20.26) | 7.25 (14.06)
  Chest pain: C10 D1 (n=17, 20) | 13.72 (16.91) | 8.33 (18.34)
  Chest pain: C11 D1 (n=15, 19) | 24.44 (29.46) | 7.02 (13.96)
  Chest pain: C12 D1 (n=10, 16) | 13.33 (17.21) | 2.08 (8.33)
  Chest pain: C13 D1 (n=7, 14) | 19.05 (26.23) | 4.76 (12.10)
  Chest pain: EOT (n=26, 37) | 30.77 (33.89) | 15.31 (24.34)
  Arm/shoulder pain: Baseline (n=56, 59) | 20.83 (27.39) | 20.34 (29.04)
  Arm/shoulder pain: C2 D1 (n=51, 53) | 20.91 (28.25) | 20.75 (24.66)
  Arm/shoulder pain: C3 D1 (n=45, 47) | 14.81 (25.18) | 5.67 (12.66)
  Arm/shoulder pain: C4 D1 (n=37, 47) | 18.92 (25.51) | 17.02 (30.19)
  Arm/shoulder pain: C5 D1 (n=33, 38) | 14.14 (26.39) | 14.91 (26.51)
  Arm/shoulder pain: C6 D1 (n=29, 33) | 16.09 (26.16) | 5.05 (12.14)
  Arm/shoulder pain: C7 D1 (n=28, 29) | 15.48 (23.10) | 14.94 (22.86)
  Arm/shoulder pain: C8 D1 (n=22, 26) | 16.67 (26.73) | 14.10 (19.26)
  Arm/shoulder pain: C9 D1 (n=18, 23) | 14.81 (23.49) | 13.04 (19.43)
  Arm/shoulder pain: C10 D1 (n=17, 20) | 13.73 (23.74) | 20.00 (27.36)
  Arm/shoulder pain: C11 D1 (n=14, 19) | 26.19 (29.75) | 15.79 (23.22)
  Arm/shoulder pain: C12 D1 (n=10, 17) | 23.33 (22.50) | 25.49 (32.34)
  Arm/shoulder pain: C13 D1 (n=8, 14) | 20.83 (24.80) | 19.05 (25.20)
  Arm/shoulder pain: EOT (n=26, 38) | 21.80 (33.92) | 23.68 (31.87)
  Other pain: Baseline (n=52, 57) | 28.85 (32.36) | 25.15 (34.09)
  Other pain: C2 D1 (n=49, 50) | 26.53 (28.85) | 32.67 (31.94)
  Other pain: C3 D1 (n=46, 47) | 34.06 (31.81) | 23.40 (31.79)
  Other pain: C4 D1 (n=36, 45) | 25.93 (27.73) | 28.15 (30.11)
  Other pain: C5 D1 (n=32, 38) | 25.00 (29.33) | 26.32 (33.02)
  Other pain: C6 D1 (n=28, 33) | 29.76 (26.20) | 27.27 (33.80)
  Other pain: C7 D1 (n=28, 28) | 32.14 (35.70) | 35.71 (36.21)
  Other pain: C8 D1 (n=22, 26) | 16.67 (28.64) | 25.64 (33.08)
  Other pain: C9 D1 (n=15, 23) | 31.11 (34.43) | 31.88 (34.05)
  Other pain: C10 D1 (n=16, 19) | 25.00 (28.55) | 22.81 (31.53)
  Other pain: C11 D1 (n=14, 18) | 42.86 (33.15) | 25.93 (33.44)
  Other pain: C12 D1 (n=10, 17) | 33.33 (27.22) | 27.45 (33.82)
  Other pain: C13 D1 (n=8, 14) | 29.17 (27.82) | 26.19 (29.75)
  Other pain: EOT (n=25, 37) | 34.67 (32.60) | 29.73 (36.67)
  Medicine for pain: Baseline (n=37, 35) | 60.36 (29.23) | 66.67 (28.01)
  Medicine for pain: C3 D1 (n=29, 24) | 65.52 (31.48) | 68.06 (31.82)
  Medicine for pain: C4 D1 (n=19, 29) | 63.16 (26.98) | 72.41 (23.69)
  Medicine for pain: C5 D1 (n=17, 22) | 70.59 (26.04) | 72.73 (22.15)
  Medicine for pain: C6 D1 (n=16, 17) | 66.67 (29.81) | 72.55 (24.25)
  Medicine for pain: C7 D1 (n=15, 14) | 75.56 (26.63) | 66.67 (29.24)
  Medicine for pain: C8 D1 (n=13, 16) | 66.67 (27.22) | 75.00 (25.82)
  Medicine for pain: C9 D1 (n=6, 14) | 72.23 (13.61) | 69.05 (20.52)
  Medicine for pain: C10 D1 (n=10, 10) | 73.34 (14.05) | 60.00 (26.30)
  Medicine for pain: C11 D1 (n=9, 9) | 48.15 (17.57) | 81.48 (17.57)
  Medicine for pain: C12 D1 (n=6, 9) | 55.56 (17.22) | 70.37 (20.03)
  Medicine for pain: C13 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Medicine for pain: EOT (n=15, 19) | 60.00 (22.54) | 66.67 (29.40)
  Medicine for pain: C2 D1 (n=30, 35) | 62.22 (22.72) | 71.43 (26.99)

8. Secondary Outcome: Percentage of Participants by Ribonucleic Acid (RNA) Expression Profile in Whole Blood
Description: RNA expression profiles of genes which were associated with tumor growth, angiogenesis and metastases were collected and correlated with efficacy.
Time Frame: Baseline, C1 D1, C1 D15, C2 D1, C3 D1, C4 D1 and C5 D1
Population: Data was not generated but sample was collected for banking and moved to a separate exploratory research database for future research.
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Circulating Endothelial Cells (CEC) in Blood: Total CEC
Description: Circulating endothelial cells (CECs) are noninvasive marker of vascular damage, remodeling, and dysfunction. Total CEC, plasma-vascular endothelial growth factor receptor-2 (pVEGFR2), VEGFR2, p-Beta-type platelet-derived growth factor receptor (pPDGFRB+) and PDGFRB+ were explored using CECs. Blood was collected to analyze effects of therapy on the number, viability/apoptotic state, and/or target activity/expression in CECs.
Time Frame: Baseline (C1 D1), C1 D15, C2 D1, C3 D1, C4 D1, C5 D1, C7 D1, C9 D1 and C11 D1
Population: ITT population: participants randomized with study drug designated according to initial randomization, regardless of whether participants received study drug or different drug. 'n': participants evaluated at specific time point for each group respectively. 'N' (Number of participants analyzed) signifies participants evaluable for the measure.
Measure: Mean (Standard Deviation); unit: Cells/milliliter (cells/mL)
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 58 | 59
Cells/milliliter (cells/mL)
  Baseline (n=39, 37) | 46815.38 (131531.755) | 16960.41 (25527.526)
  C1 D15 (n=27, 29) | 11780.15 (13127.847) | 21882.41 (67578.781)
  C2 D1 (n=32, 28) | 29229.09 (55724.997) | 40507.36 (82161.060)
  C3 D1 (n=24, 30) | 19517.50 (19793.722) | 25215.70 (42932.747)
  C4 D1 (n=20, 27) | 24556.05 (22434.011) | 41944.59 (70239.938)
  C5 D1 (n=18, 23) | 28266.22 (39480.209) | 37468.13 (82647.380)
  C7 D1 (n=11, 14) | 71770.91 (94182.032) | 36964.36 (60577.084)
  C9 D1 (n=7, 7) | 58680.00 (78138.794) | 107978.14 (206314.489)
  C11 D1 (n=6, 6) | 116620.83 (129577.280) | 120847.67 (140674.394)

10. Secondary Outcome: Circulating Endothelial Cells (CEC) in Blood
Description: as for outcome 9
Time Frame: Baseline (C1 D1), C1 D15, C2 D1, C3 D1, C4 D1, C5 D1, C7 D1, C9 D1 and C11 D1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Flourescent Intensity Unit (FIU)
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 58 | 59
Flourescent Intensity Unit (FIU)
  Baseline (pVEGFR2+) (n=50, 42) | 1936317.98 (1252665.900) | 1764577.67 (1331540.549)
  C1 D15 (pVEGFR2+) (n=38, 37) | 1822095.74 (1678888.153) | 1810049.32 (1330590.809)
  C2 D1 (pVEGFR2+) (n=41, 35) | 1767065.44 (1442193.213) | 2090673.60 (1659128.892)
  C3 D1 (pVEGFR2+) (n=33, 34) | 1715569.39 (1515661.662) | 1578940.53 (1274415.109)
  C4 D1 (pVEGFR2+) (n=25, 32) | 1472447.68 (970463.341) | 1815402.16 (1263516.725)
  C5 D1 (pVEGFR2+) (n=24, 26) | 2208801.96 (3098289.400) | 1794843.58 (1458412.725)
  C7 D1 (pVEGFR2+) (n=16, 16) | 1405048.00 (879770.893) | 1634128.00 (1443612.089)
  C9 D1 (pVEGFR2+) (n=12, 11) | 2280989.75 (1050678.808) | 2283985.00 (1093158.760)
  C11 D1 (pVEGFR2+) (n=10, 9) | 1828224.90 (1179020.490) | 2354939.11 (1116283.011)
  Baseline (VEGFR2+) (n=50, 42) | 1694522.56 (1534520.504) | 1841618.36 (1300088.201)
  C1 D15 (VEGFR2+) (n=38, 37) | 1634956.89 (1285333.248) | 1740268.05 (1444881.394)
  C2 D1 (VEGFR2+) (n=41, 35) | 1597041.59 (865675.123) | 1444404.94 (1097875.465)
  C3 D1 (VEGFR2+) (n=33, 34) | 1443986.61 (843071.909) | 1504595.71 (1163469.112)
  C4 D1 (VEGFR2+) (n=25, 32) | 1181666.88 (673860.407) | 1259913.44 (765707.741)
  C5 D1 (VEGFR2+) (n=24, 25) | 1371956.00 (948166.942) | 1447188.88 (885864.695)
  C7 D1 (VEGFR2+) (n=16, 16) | 1028231.44 (495059.378) | 1317560.13 (720095.027)
  C9 D1 (VEGFR2+) (n=12, 11) | 1485819.58 (953884.288) | 1476621.00 (1688887.819)
  C11 D1 (VEGFR2+) (n=10, 9) | 1573298.80 (1152155.993) | 1332064.78 (668964.428)
  Baseline (pPDGFRB+) (n=50, 42) | 1646702.34 (1482336.244) | 1734853.24 (1485338.326)
  C1 D15 (pPDGFRB+) (n=38, 37) | 1253893.97 (894629.298) | 1599671.65 (1669690.889)
  C2 D1 (pPDGFRB+) (n=41, 35) | 1395311.88 (1111766.454) | 1885684.31 (1356916.305)
  C3 D1 (pPDGFRB+) (n=33, 34) | 1470448.94 (841336.398) | 1285439.44 (1083860.541)
  C4 D1 (pPDGFRB+) (n=25, 32) | 1046445.72 (588769.375) | 1514713.97 (1150805.007)
  C5 D1 (pPDGFRB+) (n=24, 26) | 2253114.67 (3314986.569) | 2299459.38 (5140939.706)
  C7 D1 (pPDGFRB+) (n=16, 16) | 1380133.19 (1002147.826) | 2163313.88 (3720352.717)
  C9 D1 (pPDGFRB+) (n=12, 11) | 2172539.75 (2323386.087) | 2225289.18 (1126401.528)
  C11 D1 (pPDGFRB+) (n=10, 9) | 1580028.90 (927582.364) | 3127640.22 (2817719.865)
  Baseline (PDGFRB+) (n=50, 42) | 1775826.12 (1485762.540) | 3176459.69 (3222201.986)
  C1 D15 (PDGFRB+) (n=38, 37) | 1589914.37 (985828.939) | 1819988.05 (1807664.991)
  C2 D1 (PDGFRB+) (n=41, 35) | 1840677.73 (1315688.806) | 1586256.17 (1092406.544)
  C3 D1 (PDGFRB+) (n=33, 34) | 1690163.33 (1064816.034) | 1518360.71 (1286285.813)
  C4 D1 (PDGFRB+) (n=25, 32) | 1288624.64 (641546.254) | 1408366.91 (1013859.813)
  C5 D1 (PDGFRB+) (n=24, 26) | 1309639.50 (975890.557) | 1364500.50 (1058758.211)
  C7 D1 (PDGFRB+) (n=16, 16) | 1049351.00 (587546.139) | 1287039.25 (922009.811)
  C9 D1 (PDGFRB+) (n=12, 11) | 1666413.67 (1465165.325) | 1625161.64 (1467355.491)
  C11 D1 (PDGFRB+) (n=10, 9) | 1533606.00 (1258733.501) | 1959067.11 (1973194.943)

11. Secondary Outcome: Plasma Concentration of Soluble Proteins
Description: Plasma concentrations of soluble proteins (soluble- stem-cell factor receptor (sKIT) vascular endothelial growth factor [VEGF], and vascular endothelial growth factor receptor-2 [VEGFR2], VEGFR3) may be associated with tumor angiogenesis or tumor physiology and may correlate with efficacy or biological activity. It is presented as ratio to baseline, which is obtained by dividing the plasma soluble protein concentration at each time point by its concentration at baseline.
Time Frame: Baseline, C1D1, C1D15, C2D1, C3D1, C4D1, C5D1, C7D1, C9D1 and C11D1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Picogram/mL (pg/mL)
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 57 | 58
Picogram/mL (pg/mL)
  Baseline (SKIT) (n=52, 47) | 49740.29 (16998.69) | 49544.15 (14803.62)
  C1 D15 (SKIT) (n=42, 36) | 53095.48 (18233.85) | 55801.39 (22058.63)
  C2 D1 (SKIT) (n=41, 43) | 52979.39 (18018.73) | 55729.65 (21476.66)
  C3 D1 (SKIT) (n=40, 38) | 53817.75 (19638.72) | 65634.14 (27097.91)
  C4 D1 (SKIT) (n=32, 38) | 56961.41 (20828.07) | 72671.32 (33207.22)
  C5 D1 (SKIT) (n=27, 34) | 58305.00 (20311.85) | 68677.21 (30073.83)
  C7 D1 (SKIT) (n=18, 23) | 50701.11 (17927.98) | 75547.61 (24458.54)
  C9 D1 (SKIT) (n=12, 16) | 48680.42 (14791.32) | 65990.78 (17003.08)
  C11 D1 (SKIT) (n=11, 13) | 49251.82 (19469.45) | 66920.38 (12261.25)
  Baseline (VEGF) (n=50, 48) | 95.14 (66.60) | 121.83 (141.22)
  C1 D15 (VEGF) (n=40, 37) | 117.08 (98.05) | 287.19 (171.77)
  C2 D1 (VEGF) (n=39, 43) | 127.46 (128.06) | 324.33 (153.65)
  C3 D1 (VEGF) (n=39, 38) | 148.06 (159.80) | 368.23 (151.20)
  C4 D1 (VEGF) (n=30, 38) | 197.16 (282.49) | 405.13 (173.86)
  C5 D1 (VEGF) (n=25, 34) | 184.77 (175.32) | 400.16 (165.69)
  C7 D1 (VEGF) (n=18, 23) | 226.62 (202.53) | 433.30 (172.14)
  C9 D1 (VEGF) (n=12, 16) | 273.17 (207.22) | 422.38 (157.76)
  C11 D1 (VEGF) (n=11, 13) | 339.86 (303.71) | 449.92 (144.50)
  Baseline (VEGFR2) (n=52, 48) | 9587.31 (1570.27) | 9995.00 (2185.61)
  C1 D15 (VEGFR2) (n=42, 37) | 7828.10 (1959.39) | 10781.35 (2311.90)
  C2 D1 (VEGFR2) (n=41, 43) | 7477.80 (2146.89) | 10330.00 (2511.23)
  C3 D1 (VEGFR2) (n=40, 38) | 7058.50 (2037.12) | 10129.47 (2244.65)
  C4 D1 (VEGFR2) (n=32, 38) | 6885.94 (1754.19) | 9934.21 (1785.78)
  C5 D1 (VEGFR2) (n=27, 34) | 6565.93 (1755.75) | 10140.59 (2056.40)
  C7 D1 (VEGFR2) (n=18, 23) | 6401.11 (2360.24) | 10339.57 (1897.95)
  C9 D1 (VEGFR2) (n=12, 16) | 6291.67 (2235.24) | 9421.25 (2446.42)
  C11 D1 (VEGFR2) (n=11, 13) | 5696.36 (2724.57) | 9222.31 (2727.04)
  Baseline (VEGFR3) (n=52, 48) | 44390.77 (75118.17) | 24718.33 (12494.07)
  C1 D15 (VEGFR3) (n=42, 37) | 33684.29 (52617.02) | 17693.51 (9679.53)
  C2 D1 (VEGFR3) (n=41, 43) | 35780.49 (68287.68) | 17798.37 (9710.23)
  C3 D1 (VEGFR3) (n=40, 38) | 34147.00 (74220.30) | 15901.32 (8062.41)
  C4 D1 (VEGFR3) (n=32, 38) | 19730.94 (9237.69) | 16307.37 (7409.61)
  C5 D1 (VEGFR3) (n=27, 34) | 17452.59 (8614.99) | 16381.47 (6707.41)
  C7 D1 (VEGFR3) (n=18, 23) | 17896.67 (8360.82) | 15626.30 (8873.31)
  C9 D1 (VEGFR3) (n=12, 16) | 21449.17 (12806.75) | 14733.44 (6441.61)
  C11 D1 (VEGFR3) (n=11, 13) | 22332.73 (12408.37) | 16048.46 (7064.47)

12. Other Pre Specified Outcome: Plasma Concentration Change in the Uridine Diphosphate Glucuronosyltransferase 1A1 (UGT1A1) Genotype
Description: UGT1A1 an enzyme of the glucuronidation pathway that transforms small lipophilic molecules, such as steroids, bilirubin, hormones, and drugs, into water-soluble, excretable metabolites.
Time Frame: Baseline (Day 1 of Cycle 1)
Population: Data was reported in listings but not summarized due to statistical constraints.
Groups:
- Bevacizumab+ Paclitaxel + Carboplatin: Axitinib (AG-013736) 5 mg tablet administered orally BID along with IV infusion of paclitaxel 200 mg per square meter (mg/m^2) over 3 hours and carboplatin AUC of 6 mg*min/mL infusion over 30 minutes in cycles of 3 weeks. After completion or discontinuation of treatment for reasons other than disease progression, participants continued to receive Axitinib (AG-013736) BID maintenance therapy.
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab+ Paclitaxel + Carboplatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib + Paclitaxel + Carboplatin | Bevacizumab + Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 31/58 | 19/59
Other Adverse Events (participants affected / at risk) | 54/58 | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Paclitaxel + Carboplatin (N=58) | Bevacizumab + Paclitaxel + Carboplatin (N=59)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 3 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 7 | 3
Fatigue (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Meningeal disorder (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Paclitaxel + Carboplatin (N=58) | Bevacizumab + Paclitaxel + Carboplatin (N=59)
Anaemia (Blood and lymphatic system disorders) | 12 | 15
Leukopenia (Blood and lymphatic system disorders) | 7 | 5
Neutropenia (Blood and lymphatic system disorders) | 18 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 11
Hypothyroidism (Endocrine disorders) | 9 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 16 | 17
Diarrhoea (Gastrointestinal disorders) | 27 | 20
Dyspepsia (Gastrointestinal disorders) | 8 | 2
Nausea (Gastrointestinal disorders) | 21 | 19
Stomatitis (Gastrointestinal disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 14 | 11
Asthenia (General disorders) | 17 | 6
Chest pain (General disorders) | 8 | 3
Fatigue (General disorders) | 20 | 22
Malaise (General disorders) | 3 | 0
Mucosal inflammation (General disorders) | 5 | 3
Pain (General disorders) | 6 | 6
Pyrexia (General disorders) | 6 | 9
Lower respiratory tract infection (Infections and infestations) | 4 | 6
Urinary tract infection (Infections and infestations) | 4 | 3
Weight decreased (Investigations) | 10 | 6
Decreased appetite (Metabolism and nutrition disorders) | 25 | 12
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 10
Dizziness (Nervous system disorders) | 5 | 4
Dysgeusia (Nervous system disorders) | 4 | 6
Headache (Nervous system disorders) | 11 | 4
Lethargy (Nervous system disorders) | 4 | 5
Neuropathy peripheral (Nervous system disorders) | 15 | 15
Paraesthesia (Nervous system disorders) | 6 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Polyneuropathy (Nervous system disorders) | 3 | 2
Syncope (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 4 | 4
Depression (Psychiatric disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 10 | 8
Proteinuria (Renal and urinary disorders) | 6 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 27
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 6
Hypertension (Vascular disorders) | 24 | 25
Hypotension (Vascular disorders) | 6 | 1
Oedema peripheral (General disorders) | 2 | 6
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 3
Respiratory tract infection (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Neurotoxicity (Nervous system disorders) | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.